## **Evaluation of SkillTalk for Autistic Young Adults**

Informed Consent Form NCT06281171 September 29, 2023

# Consent to Participate in Evaluation Study of SkillFlix for Autistic Young Adults

#### What is this about?

We are creating an online resource library for young adults on the autism spectrum. The resource is about healthy relationships, and other important areas of life, like coping with stress, employment, and advocacy. We want to see if the online resource library helps people communicate.

If you take part in this study, you may be asked to use this online resource library. You will be asked to complete three online surveys and do roleplays with a research team member of your choice. This will help us learn whether the online resource library was helpful for you.

#### Who are we?

We are from dfusion, a small business that makes products to improve health. dfusion has done many research studies with youth and adults. This project is funded by the National Institute on Disability, Independent Living, and Rehabilitation Research.

#### What would I be asked to do?

We will divide the participants into two groups. There is a fifty-fifty chance to be in either group. You will either be in the video library group or in the online flyer group. The video library group will watch the videos right away. The online flyer group will wait four months to watch the videos, if they choose.

#### Regardless of group, all participants will be asked to:

- Do a role-play with a study team member of your choice. The role-plays are brief, happen over Zoom, and will be recorded. This will take about 20 minutes.
- Fill out the first online survey about yourself. This will take around 30 minutes.
- Use the study materials for a month.
- After the first month of the study, you will take a second online survey and do another roleplay.
- Four months into study, you will take the final online survey and role-play.

All of these study activities will take place over 4 months and will take 4–6 hours of time or less to complete. For the each of the first two survey and roleplay events, you will receive a gift card for \$50, and for the final you will receive a gift card for \$100. You can earn up to a total of \$200 by the end of the study.

#### Are there any risks?

You may feel some discomfort answering survey questions about your relationship skills. You may feel awkward doing the roleplay scenes with study team members. To help with this, we will give you the choice to talk to one of three team members. We will send a website with pictures and a few sentences describing each person ahead of time.

The research team will keep the information you share with us confidential, including the roleplay recordings and survey information. We will replace your name with confidential identification numbers so that the information you share is not linked to your identity. A codebook that states which confidential identification number belongs with your name will be stored separately from any information you share. This codebook will be destroyed three years after the study is complete. Video files from the role play sessions will be destroyed three years after the study is complete. The information you share will not be shared with any organizations you may be affiliated with or anyone else outside of the study team with for any reason.

#### Do I have to take part?

No. You can choose whether or not to take part. Participation is voluntary and you may choose to stop participating in the study at any time with no consequences. You do not have to answer any survey questions if you do not want to. If you feel uncomfortable or distressed during the roleplay scenes, you can stop at any time.

#### Are there any costs involved?

No. There are no costs to take part in this study.

#### What are the benefits of taking part?

By taking part in this study, you will help us make sure that the online resource library is helpful and will help us improve this tool in order to support autistic people. You will have the opportunity to access new resources that may improve your relationship skills.

#### What if I have questions?

Here are two people you can call for more details about the project:

Lane Edwards, Project Director: (303)862-1957; lane.edwards@dfusioninc.com

Rachel Firpo, Research Assistant: (925)234-5746; rachel.firpo@dfusioninc.com

Confidentiality is not guaranteed when using email.

For questions about your rights as a participant in this research project call:

Dr. Tanya Matthews, IRB Chairperson: (866) 537-5030. An IRB is a committee that helps to make sure people in research projects are protected.

#### How do I give consent for myself to take part?

We need your written consent before you can take part in the study. Please complete the consent form on the following page to indicate your decision (yes or no) to participate in the study. You can only participate if you answer "YES". We are happy to answer any questions you have about the study before you decide whether or not to consent to participate. We will also ask you several questions to make sure you understand the study.

Thank you.

## Consent to Participate in Evaluation Study of SkillFlix for Autistic Young Adults

Study Principal Investigator: Regina Firpo-Triplett, MPH

### **Participant Consent**

| Please check one box: YES—I agree to take part in the research this form describe | es. |
|---|---|
| □ NO—I do NOT agree to take part in the research this form of | describes. |
| Please check one box about future studies: | |
| ☐ YES—I would like to be contacted about future research s | studies. |
| ☐ NO—I do NOT want to be contacted about future research | ch studies. |
| If you checked YES for either of the above, please print and sign yo provide the best contact information for you. | our name, fill in the date, and |
| Your Name: | |
| Date: | |
| Phone Number: | |
| Email: | |
| If under guardianship or conservatorship, please attain a consent sign | gnature from your guardian. |
| Guardian's Name: | |
| Guardian's Signature: | Date: |

### **Consent Comprehension Questions and Protocol**

Instructions for Staff: The staff person conducting the consent protocol will ask the following questions and note whether the potential participant provides a correct answer or needs to be corrected. If the staff person is unsure, go on to the next question and come back to that question. People do not need to answer questions correctly on the first trial. However, they need to show comprehension on all questions after being corrected to be able to participate in the study. People who are not able to engage with this task (e.g., answering questions when asked) are not able to participate in the study.

Say, "I would like to ask you some questions to make sure you understand what you are agreeing to."

- 1) We are making a video library. What will the video library help people do?
  - a. A correct answer will include references to (a) learning skills, getting better at, and (b) relationships, employment, coping with stress, self-advocacy.
- 2) What are a couple of the things that we will ask you to do as part of the study?
  - a. A correct answer will include at least one of the following: (a) filling out online surveys, (b) watching videos from the online video library, OR some will be asked to watch videos now, some later/in 4 months, and (c) taking part in roleplay scenarios.
- 3) Are there any risks in participating in the study?
  - a. A correct answer will include reference to feeling awkward or uncomfortable answering questions on the survey or participating in the roleplays.
- 4) Do you have to participate in the study?
  - a. The correct answer is no, they do not have to participate in the study.

**NOT ELIGIBLE MESSAGE:** Thank you for answering my questions. Based on our conversation, you are not eligible to participate in this study, but please let me know if you would like us to contact you about future studies for which you may be eligible.

**ELIGIBLE MESSAGE:** Thank you for answering my questions. Based on our conversation, you are eligible to participate in the study.

| Question 1 | |
|---|---|
| ☐ Correct | Question 3 |
| ☐ Understood with correction | ☐ Correct |
| ☐ Incorrect after correction | <ul> <li>Understood with correction</li> </ul> |
| ☐ Did not answer | <ul><li>Incorrect after correction</li></ul> |
| | ☐ Did not answer |
| Question 2 | |
| ☐ Correct | Question 4 |
| <ul><li>Understood with correction</li></ul> | ☐ Correct |
| ☐ Incorrect after correction | <ul> <li>Understood with correction</li> </ul> |
| ☐ Did not answer | <ul><li>Incorrect after correction</li></ul> |
| | ☐ Did not answer |